CLINICAL TRIAL: NCT00006389
Title: A Phase II Combination Trial of Bryostatin-1 and Cisplatin in the Treatment of Metastatic Gastric Cancer
Brief Title: Bryostatin 1 and Cisplatin in Treating Patients With Metastatic or Unresectable Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02361; NCI-2012-02361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CHNMC-PHII-22; CDR0000068267; NCI-T99-0040; PHII-22 (USC 3S-00-1) (Other: University of Southern California); T99-0040 (Other: CTEP); N01CM17101 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2013-10

CONDITIONS: Stage III Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — bryostatin 1; Bryostatins; Cisplatin

ARMS (1):
- Treatment (Experimental): Patients receive bryostatin 1 IV over 72 hours on days 1-3 followed by cisplatin IV over 1 hour on day 4. Treatment repeats every 3 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bryostatin 1; Drug: cisplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bryostatin 1 — Given IV
  Other Names: B705008K112; BRYO; Bryostatin
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of bryostatin 1 and cisplatin in treating patients who have metastatic or unresectable stomach cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bryostatin 1 may increase the effectiveness of cisplatin by making tumor cells more sensitive to the drug. Combining cisplatin with bryostatin 1 may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate and survival in patients with metastatic or unresectable carcinoma of the stomach treated with bryostatin 1 and cisplatin.

II. Determine the toxic effects of this regimen in these patients. III. Determine the molecular determinants of response to this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive bryostatin 1 IV over 72 hours on days 1-3 followed by cisplatin IV over 1 hour on day 4. Treatment repeats every 3 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic or unresectable carcinoma of the stomach
* Measurable disease
* No brain metastasis
* Performance status - Karnofsky 70-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* No history of any bleeding disorders
* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2 times normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No history of peptic ulceration or gastrointestinal bleeding
* No active infection
* No seizure disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other serious concurrent illness that would preclude study entry
* No medical, social, or psychological factors that would preclude study entry
* No prior chemotherapy
* No prior radiotherapy
* More than 4 weeks since prior major surgery
* Prior incomplete resection allowed
* No other prior antitumor treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2000 through March 2002, a total of 12 patients signed a consent form and were enrolled on this study: 2 from COH, 8 from USC and 2 from UCD. All patients received treatment.
Groups:
- Treatment: Patients received byrostatin-1 45µg/m2/day as a 72 hour intravenous infusion followed by a 1-hour infusion of cisplatin 50 mg/m2 on day 4 immediately at the bryostatin-1 infusion, administered every three weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.
  bryostatin 1: Given IV
  cisplatin: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Observed Response Rate.
Description: All patients had measurable disease and were assessed after 2 cycles of chemotherapy by medical photograph, plain x-ray, CT, MRI or other imaging scans of at least 2.0 cm or greater with conventional techniques or 1.0 cm or greater with spiral CT. Patients were evaluated by RECIST criteria. All measurable lesions, up to 10 "target lesions" were recorded and measured at baseline across the longest diameter (LD). All other non-target lesions were documented as present or absent. Complete Response (CR) was defined as complete disappearance of the tumor, partial response (PR) was defined as at least a 30% decrease of the sum of the LD of the target lesions, using the baseline sum LD as the reference
  The observed response rate was defined as the percentage of evaluable patients whose best response is a CR or PR with associated 95% confidence interval.
Time Frame: Best response recorded from the start of treatment until disease progression/recurrence. Assessed every 2 cycles.
Population: The first 15 patients accrued to an Optimal Three-Stage Phase II design. If 3 or more responses are seen then 18 additional evaluable patients will be accrued to the second stage.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Percentage of Participants | 0 [0 to 26.5]

2. Secondary Outcome: Overall Survival
Description: Overall survival was estimated according to the Kaplan-Meier product-limit method.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment
Number analyzed (Participants) | 12
Months | 2.7 [1.6 to 5.3]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was estimated according to the Kaplan-Meier product-limit method
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 12
months | 1.2 [1.0 to 2.2]

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: All adverse events (all grades & attributions) that were not identified as serious are included in "Other" events table.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 10 (20)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 8 (15)
Vomiting (Gastrointestinal disorders) | 8 (12)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1 (1)
Edema (General disorders) | 5 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (17)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2)
Rigors/chills (General disorders) | 1 (1)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 (6)
Alkaline phosphatase (Investigations) | 6 (8)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (2)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1)
Creatinine (Investigations) | 3 (5)
FEV(1) (Investigations) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Leukocytes (total WBC) (Investigations) | 4 (7)
Lymphopenia (Investigations) | 8 (14)
Neutrophils/granulocytes (ANC/AGC) for leukemia studies or bm infiltrative/myelophthisic (Investigations) | 1 (1)
Platelets (Investigations) | 4 (9)
Weight loss (Investigations) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (15)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (6)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 (10)
Dizziness (Nervous system disorders) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 3 (5)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Pain (Nervous system disorders) | 9 (29)
Confusion (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Mood alteration (Psychiatric disorders) | 3 (3)
Obstruction, GU (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Of 12 pts accrued\treated, none responded. The initial phase accrual goal was 15, but given the 12 non-responders, we determined the probability of 3 future pts all responding (stochastic curtailed sampling) at 2.7%. Decided to terminate the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less